CLINICAL TRIAL: NCT03991390
Title: Effectiveness of Visual Feedback Laser and Core Stability Exercises for Balance Impairment in Subacute Stroke Patients With Pusher Syndrome
Brief Title: Effectiveness of Balance Exercise Program for Stroke Patients With Pusher Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Parc Sanitari Pere Virgili (Other)
Collaborators: Universitat Internacional de Catalunya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pusher Syndrome - PSPV
Record Dates: First submitted 2019-06-12; First posted 2019-06-19 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Pusher Syndrome; Subacute Stroke
Keywords: Pusher syndrome; Core stability; Visual feedback; Postural control; Balance; Rehabilitation stroke
MeSH Terms: interventions — Feedback, Sensory

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Core stability and feedback visual laser exercises (Experimental): Two complementary protocols for the treatment of balance after stroke in patients with pusher syndrome were designed, including multidimensional physiotherapy exercises. Both protocols differentiate 3 levels of difficulty: Second level requires maintenance of balance sitting 5", if the patient does not succeed, stays in level 1. To move to L3 patients must stay seated 10''. Each exercise is repeated 5 times, always considering patients' levels of fatigue and safety.
  Visual feedback with laser (Motion Guidance Clinical Kit, approved for therapeutic use): Through visual aid, patients' verticality is achieved by encouraging their active participation in correcting the imbalance while performing the exercises.
  Core stability: The exercises have to be adapted for the pusher patient avoiding overuse of the less affected side of the body, and strengthening the muscles that stabilize the trunk.
  Interventions: Other: Visual Feedback and Core Stability exercises protocol
- Control stroke (Active Comparator): Rehabilitation program is based on a comprehensive approach, where the patient follows a personalized plan of exercises according to the deficits, the previous situation and personal concerns.
  Interventions: Other: Control stroke

INTERVENTIONS:
Other: Visual Feedback and Core Stability exercises protocol — This arm consists of 5 sessions per week, 60 minutes each. One session consists of 30 minutes of conventional physiotherapy and 30 minutes of Core Stability exercises and laser visual feedback exercises, on alternate days.
  All sessions will be performed by the same physiotherapist.
  Arms: Core stability and feedback visual laser exercises
Other: Control stroke — This arm consists of 5 sessions per week, 60 minutes each comprising usual physiotherapy treatment.
  All sessions will be performed by the same physiotherapist.
  Arms: Control stroke

SUMMARY:
The objective of this study is to evaluate whether the application of two laser visual feedback exercises and core stability exercises can positively influence postural orientation and the perception of postural verticalization compared to conventional treatments, with the final goal of improving the balance in sitting and standing and the functionality in activities of daily living.

DETAILED DESCRIPTION:
Study designed as a randomized clinical trial. The total sample (N=16) will randomized into two groups: treatment vs. control. All of them suffering from subacute stroke and pusher syndrome.

The study intervention will last 4 weeks. The control group will receive usual rehabilitation treatment for patients with stroke and pusher syndrome (60 minutes per day/5 days per week). The intervention group will receive usual rehabilitation treatment for patients with stroke and pusher syndrome (30 minutes per day/5 days per week) plus 30 minutes of therapy based on the specific protocol designed for the study. This protocol will consist of Core Stability exercises and visual feedback with lasers, both procedures will be alternated one day each.

The evaluation of the intervention program will be based on the established objectives, assessing: 1) Pushing Intensity (controversial push scale (SCP)), 2) Laterality (Burke Scale (BLS)), 3) Balance (Postural Assessment Scale for Stroke Patients (S-PASS)), 4) patient functional capacity (Barthel Index), and 5) Quality of Life (Newcastle Stroke-Specific Quality of Life Measure (NEWSQOL)). These variables will be evaluated baseline and post-intervention. Additionally, SCP, BLS and S-PASS will be assessed 15 days after starting treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years admitted to an intermediate care unit after suffering from subacute stroke, for functional recovery.
* Diagnosis of ischemic or hemorrhagic stroke confirmed by Magnetic Resonance Imaging (MRI) or Computed Tomography (CT) scan.
* Pusher syndrome identified by the Scale for Contraversive Pushing (SCP) with a score of ≥2 and by Burke Lateropulsion Scale (BLS) with a value of ≥3.

Exclusion Criteria:

* Patients with severe previous functional dependence (Barthel Index ≤60)
* Patients diagnosed with dementia GDS-4 or previous severe cognitive impairment.
* Patients diagnosed with delirium.
* Patients diagnosed with Wernicke's aphasia.
* Patients with a previous severe visual deficit that prevents them from continuing activity (retinopathy, cataracts, etc.)
* Patient with a history of other causes of balance impairment.
* Patients with orthopedic conditions that difficult the performance of the proposed rehabilitation treatment.
* Patients enrolled in other research studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Change of Contraversive Pushing at 30 days | Baseline (admission), 15 days, 30 days
  The Scale for Contraversive Pushing (SCP) allows to diagnose and quantify the pushing behavior of the post-stroke patient. This scale is based on the three main signs of pusher behavior:
  * Symmetry of the spontaneous posture,
  * Push of the upper or lower non-affected limb towards the affected side,
  * Resistance to a passive correction of posture,
  Assigning up to 1 point in each subscale and in each position. The maximum score is 6, this being the maximum expression of the pusher behavior.
Change of Lateropulsion at 30 days | Baseline (admission), 15 days, 30 days
  The Burke Lateropulsion Scale (BLS) is a complementary scale appropriate to the "Contraversive Pushing" scale in the follow-up of patients with pusher behavior in relation to the resistance to passive correction shown by the patient in supine, turning, sitting, standing, walking and transfers scoring up to 17 points.
  The scale evaluates the patient in sitting and standing position. The patient will be tilted 30º to the affected side and will be asked to return to the vertical position, according to the degrees where resistance appears will be given a score (0 there is no resistance, 1 resistance that begins at 5º, 2 the resistance begins at 10º, 3 the resistance begins above 10º) and the examiner will score if it is (0-null,1-light, 2-moderate, 3-severe) and the same will be evaluated when standing.
  Interobserver reliability has been shown to be effective for therapy.
Change of Balance at 30 days | Baseline (admission), 30 days
  The S-PASS scale has been validated for post-stroke patients in Spanish. It consists of 12 items and is subdivided into two: mobility (7 items) and balance (5 items). The total score of the scale is 36 points and the score goes from 0 to 3 on each item. The scale also quantifies the help the patient needs to perform each action.
  In items 1 to 4 and 8, control of the trunk is evaluated, both on the affected side and on the non-affected side. Items 5 to 7 report anticipatory postural adjustments, in transfers. Items 9 and 10 assess the balance in standing with and without help, respectively, and finally, on items 11 and 12, the one-leg support in affected and not affected leg without help.

SECONDARY OUTCOMES:
Change of Quality of Life at 30 days | Baseline (admission), 30 days
  The Newcastle Stroke-Specific Quality of Life Measure (NEWSQOL) assesses quality of life in patients suffering from ischemic or hemorrhagic stroke.
  The questionnaire consists of 56 items distributed in 11 domains: mobility, activities of daily living, pain, vision, cognition, communication, feelings, interpersonal relationships, emotions, sleep and fatigue. In each item the commentary 'due to stroke' is added to differentiate the specific impact of the stroke from other health or social problems, or from natural aging process.
  Each item is scored on 4 points (0 to 3). The domain scores are obtained by adding the results of the items included in that domain and then adding each domain to achieve a final score. Higher scores indicate a greater impact on the quality of life of the individual.
  The time is difficult to calculate according to the patient's condition can range between 30 and 45 minutes
Change of Independence in the basic activities of daily life at 30 days | Baseline (admission), 30 days
  Measured by the Barthel Index. The Barthel index is a questionnaire with 10 items that assesses the independence of the development of basic activities of daily life (eating, washing, dressing, arranging, evacuating, urinating, going to the toilet, mobile chair, walking and climbing and going down stairs) . The score ranges from 0-100, total dependence, Maximum independence. More specifically, the results are classified as follows: <20 total dependence, 21-60 severe dependence, 61-90 moderate dependence, 91-99 slight dependence, 100 independence.

CONTACTS AND LOCATIONS:
Overall Officials: Caritat Bagur, PhD, Study Director — Universitat Internacional de Catalunya
Locations (1):
- Parc Sanitari Pere Virgili, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No